CLINICAL TRIAL: NCT02536612
Title: Empower, Nudge: Increasing Dual Protection Among Young Women in South Africa
Brief Title: Empower, Nudge: Increasing Dual Protection in South Africa
Acronym: EN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Omar Galarraga, PhD, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIA14-68
Record Dates: First submitted 2015-08-20; First posted 2015-09-01 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: HIV; Pregnancy; STDs
Keywords: Motivation; Behavioral Economics; Conditional Economic Incentives; Conditional cash transfers; Contingency management
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lottery (Experimental): Conditional economic incentive (CEI) lotto arm participants will get a chance to win a type of lottery or "lotto" ticket with a 50% chance of winning each time: (a) if they come back to the clinic and are still using a modern contraception method after 3 months (including IUD, injectable contraceptive, or implant); (b) if they come back to the clinic and are still using modern contraception after 6 months; and (c) if they come back to the clinic at 6 months and they don't have a new curable STD (such as syphilis).
  They will also will receive reimbursement to cover their transport and time at baseline, at 3 months and at 6 months.
  Interventions: Other: Lottery
- No Lottery (Active Comparator): Participants in the Control (No CEI Lotto) group will receive reimbursement to cover their transport and time at baseline, at 3 months and at 6 months; they will NOT have a chance to win a lottery even if they are still using a modern contraception and are free of new curable STDs.
  Interventions: Other: No Lottery

INTERVENTIONS:
Other: Lottery — Opportunity for entry in lottery (each time, at months 3 and 6).
  Other Names: Lotto; Empower Lotto Bowl
  Arms: Lottery
Other: No Lottery — Transport compensation for study visits at baseline and at months 3 and 6. No chance to win lottery ticket.
  Arms: No Lottery

SUMMARY:
The purpose of the study is to test feasibility and acceptability of a lottery to help women in Cape Town, South Africa to continue using long-acting reversible contraceptives to avoid unintended pregnancies, and to also use condoms to reduce sexually transmitted infections including HIV.

DETAILED DESCRIPTION:
The overall objective is to implement a pilot project offering conditional economic incentives (CEI) for dual protection (the prevention of HIV or other sexually transmitted infections and pregnancy via the simultaneous use of condoms plus effective contraception) among young women in Cape Town, South Africa, to test feasibility and acceptability, and to gather preliminary evidence on effect sizes to inform a future efficacy trial. CEI are an innovative structural approach for dual protection, which so far has not been tested in generalized HIV epidemic settings. The project has three aims. First, it will test the feasibility and acceptability of a conditional economic incentive (CEI) program to incentivize dual protection among young women in Cape Town. The working hypothesis is that a program with modest economic incentives in the form of a lottery to continue using modern contraception and stay free of sexually transmitted infections (STI) can be implemented among young women who express a desire to avoid unintended pregnancies. The hypothesis is that the CEI treatment group will exhibit greater program participation and retention rates as compared to the control group. Second, the study will obtain estimates of the effect of CEI on the primary outcomes (adherence to the dual protection regimen) through: (1) continuation of a contraceptive method of choice throughout the six month study period, and (2) self-reported condom use. Contraceptive continuation will be measured via clinic records (proxy for clinical checkup) at the 3 and 6 month follow up visits. Self-reported condom use will not be used to provide any incentives. The hypothesis is that receipt of CEI (lotteries) will be associated with higher rates of dual protection. Third, the study will examine the degree to which CEI (lotteries) impact secondary outcomes: a urine pregnancy test and STI status (measured at baseline and 6 month follow up). A selected STI (syphilis) will be monitored for assessment of the STI outcome, using a rapid test that can be administered at clinic level. The working hypothesis is that the participants in the CEI (lottery) treatment group will have reduced rates of STI and they will have lower rates of pregnancy.

This pilot trial will include young women, ages 18-40, recruited from a community clinic in Cape Town. A maximum of 96 women will be randomly assigned to one of two arms (n=48 each) in a randomized controlled trial design. In the trial, Arm 1 (control) will receive transport compensation for study visits at each of the study visits at baseline and at months 3 and 6. Arm 2 (intervention) will receive transport compensation for study visits at each visit at baseline and at months 3 and 6, plus the opportunity for entry in a lottery. Participants in Arm 2 will have a chance to receive two lottery tickets: (a) the first when returning by month 3, subject to confirmation of continued use of the participant's preferred contraceptive; (b) the second upon completion of the six month study period, subject to confirmation of continued use of the participant's preferred contraceptive over the course of the 6 month study period; and if they are free of a new curable STI. The lottery tickets will enter the participant into a drawing for a prize at month 3 and at the end of the six month study period. All participants will receive transport compensation each time at baseline, month 3 and month 6. There will be 15-20 minute follow-up sessions for everyone at months 3 and 6 when receiving STI results, and CEI (lotteries) for those in the treatment group. At month 3, follow-up sessions will include some reinforcement of key messages related to dual protection. At months 3 and 6, the follow-up sessions will include administration of the study questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ages 18-40 years
* Has been pregnant within the last 12 months (and has either delivered a baby, had a miscarriage, or an abortion within the last 12 months).
* Has chosen one of the following contraceptive methods: IUD, Implant, or injectable

Exclusion Criteria:

* Unwillingness to sign an informed consent to participate in research
* Unwillingness to participate in the Control group, if so assigned in the randomization

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Retention in the study | 6 months

SECONDARY OUTCOMES:
Long-acting contraceptive continuation | 6 months
  continuation of a contraceptive method of choice throughout the six month study period
Condom use | 6 months
  Self-reported condom use (male and/or female)

OTHER OUTCOMES:
Combined composite STDs | 6 months
  Composite STDs (syphilis and HIV)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Galarraga, PhD, Principal Investigator — Brown University School of Public Health; Abigail Harrison, PhD, Principal Investigator — Brown University School of Public Health; Jane Harries, PhD, Study Director — University of Cape Town
Locations (1):
- Lady Michaelis Community Health Clinic, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Galarraga O, Harries J, Maughan-Brown B, Cooper D, Short SE, Lurie MN, Harrison A. The Empower Nudge lottery to increase dual protection use: a proof-of-concept randomised pilot trial in South Africa. Reprod Health Matters. 2018 Dec;26(52):1510701. doi: 10.1080/09688080.2018.1510701. PMID 30212281
- [Result] Sullivan ME, Harrison A, Harries J, Sicwebu N, Rosen RK, Galarraga O. Women's reproductive decision making and abortion experiences in Cape Town, South Africa: A qualitative study. Health Care Women Int. 2018 Nov;39(11):1163-1176. doi: 10.1080/07399332.2017.1400034. Epub 2017 Dec 15. PMID 29111909